CLINICAL TRIAL: NCT07251712
Title: A Phase I Open-label Trial in Healthy Volunteers to Evaluate the Exposure of Aramchol From Two Different Single Doses of an Aramchol Meglumine Tablet
Brief Title: Single and Multiple Dose Pharmacokinetics (PK) of Aramchol From an Aramchol Meglumine Tablet
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AM-003; 1013148 (Registry Identifier: IRAS); IRAS number- 1013148 (Other: Galmed Pharma)
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — aramchol

STUDY DESIGN:
Intervention Model Description: Each participant will attend 2 trial sessions in a crossover design with a wash-out interval of at least 14 days between dosing in each session.
Masking Description: This will be an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A- Administration of Aramchol Meglumine tablet (Experimental): 12 subjects will be randomized to Part A. Participants will receive Aramchol meglumine tablet (test formulation) at 2 different single doses and plasma concentration will be assessed.
  Interventions: Drug: Aramchol
- Part B- Administration of Aramchol meglumine or Aramchol acid tablets (Experimental): 20 subjects will be randomized to Part B. Participants will receive Aramchol meglumine once daily for 10 days based on a dose predicted in Part A. Steady-state plasma concentration of Aramchol will be assessed.
  Interventions: Drug: Aramchol

INTERVENTIONS:
Drug: Aramchol — Aramchol tablet at 2 different single doses
  Other Names: 3β-arachidylamino-7α,12α-dihydroxy-5β-cholan-24-oic acid

SUMMARY:
Evaluate the exposure of of Aramchol from 2 different single doses of Aramchol meglumine tablet and to compare the exposure of steady state from a selected dose of Aramchol meglumine tablet.

DETAILED DESCRIPTION:
Evaluate the exposure of of Aramchol from 2 different single doses of Aramchol meglumine tablet and to compare the exposure of steady state from a selected dose of Aramchol meglumine given one daily with that from a 300 mg dose of Aramchol free acid tablets given twice daily in adult Healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers with body mass index (BMI) in the range of 18-30.9 kg/ m2 inclusive
* Deemed healthy on the basis of clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine
* Agree to follow-up the contraception requirements of the trial
* Able to give fully informed written consent

Exclusion Criteria:

* Females of reproductive potential who are pregnant or lactating
* Positive tests for hepatitis B, C or HIV
* History of sever adverse reaction to any drug
* Known sensitivity to drug medication
* Drug or alcohol abuse
* Smoking in the 3 months prior the study
* Clinically relevant abnormal lab results, medical history or concurrent medical condition
* Evidence of acute or chronic disease
* Inability to adhere to study requirements

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Maximum observed peak concentration (Cmax) of Aramchol | 2 months
  Blood samples will be collected for pharmacokinetics characterization. Cmax will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Time to reach maximum concentration (Tmax) of Aramchol | 2 months
  Blood samples will be collected for pharmacokinetics characterization. Tmax will be calculated from plasma concentration-time data using non-compartmental methods based on the actual time of sample collection and summarized using descriptive statistics
Area under the plasma curve (AUC) of Aramchol | 2 months
  Blood samples will be collected for pharmacokinetics characterization. AUC of Aramchol will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.

SECONDARY OUTCOMES:
Minimum observed concentration (Cmin) of Aramchol | 2 months
  Blood samples will be collected for pharmacokinetics characterization. Cmin will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Terminal elimination half life (T1/2) of Aramchol | 2 months
  Blood samples will be collected for pharmacokinetics characterization. T1/2 will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Average observed concentration (Cavg) of Aramchol | 2 months
  Blood samples will be collected for pharmacokinetics characterization. Cavg will be calculated from plasma concentration-time data using non-compartmental methods and summarized using descriptive statistics.
Safety and tolerability of Aramchol | 2 months
  The number of participants with treatment-related adverse events, as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Christina Yeung, MBBS, Principal Investigator — HMR